CLINICAL TRIAL: NCT03489421
Title: Mitochondria in HIV and Aging (MITO+)
Acronym: (MITO+)
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2161
Record Dates: First submitted 2018-03-25; First posted 2018-04-05 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Human Immunodeficiency Virus (HIV); Mitochondrial Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV Infected
- Un-infected controls: Controls without HIV from a historical pre-approved-IRB-protocol database

SUMMARY:
Older adults with human immunodeficiency virus (HIV) and a long history of antiretroviral therapy have more mitochondrial dysfunction- the cells that help them make energy. This dysfunction in mitochondria may lead to symptoms of muscle fatigue, physical function impairment, and impaired exercise tolerance compared to HIV-uninfected controls of a similar age and body mass index (BMI). Furthermore, the investigators hypothesize that the older antiretroviral therapy (ART) of tenofovir disoproxil fumarate (TDF) is associated with greater impairment in mitochondrial function than the newer agent, tenofovir alafenamide (TAF).

ELIGIBILITY:
* Inclusion criteria:

  * Between the ages of 50-75 years at study entry (a subset of participants changing from TDF-based ART to TAF-based ART will also have mitochondrial function measured and the age range for this subset is 18-70)
  * Known HIV infection or presumed HIV uninfected (will be confirmed at screening)
  * For HIV+ participants: must be on an ART regimen (change in regimen permitted for preference/tolerability but not for virologic failure) for a minimum of 5 years, with a viral load < 200 during the prior 2 years. The investigators will initially target 10 years of therapy, but will expand to 5 years if needed for enrollment.
  * Although any ART regimen will be allowed if effective (as above), the investigators will first target participants that have a history of > 5 years of TDF exposure and are currently on TAF or TDF, but no prior exposure to AZT or stavudine.
  * CD4 T-cell count greater than 200 cells/mm3
  * All participants must be able to perform activities of daily living without assistance, and ambulate independently.
  * Sedentary as defined above
  * Post-menopausal as defined by cessation of menstrual periods for at least 12 months without any other obvious pathological or physiological cause OR removal of ovaries at least 12 months prior to enrollment.
  * Body mass index between 25-38 kg/m2
* Exclusion criteria:

  * Participation in another clinical trial where the therapy is unknown or blinded.
  * Diabetes, as defined by use of diabetes medications, hemoglobin A1c 6.5 or greater, fasting plasma glucose 126 mg/dL or greater, or random plasma glucose 200 mg/dL or greater.
  * Persons on statin therapy (as possible; this criteria may be removed for recruitment difficulties).
  * Fasting triglycerides > 400
  * Untreated or incompletely treated thyroid disease will be excluded; stable therapy for > 6 months will be allowed.
  * Persons on growth hormone or growth hormone axis therapy (i.e., tesamorelin) will be excluded.
  * The investigators will initially target men, women, or transgendered individuals without replacement hormone use. If the investigators are unable to recruit the target number of participants, stable (>3 months) estrogen or testosterone within physiologic replacement dose range will be permitted.
  * Corticosteroid use, including intra-articular, will be excluded (within 3 months for oral; within 6 months for intra-articular); inhaled or intranasal will be permitted.
  * Immunosuppressive medications within 6 months, including methotrexate, infliximab, azathioprine, etc.
  * Women that are pregnant, breast-feeding, or intend to become pregnant.
  * Known hepatitis B or C with detectable viremia within in the past 6 months.
  * Hepatitis C with undetectable viral load for at least 6 months will be allowed.
  * Known mitochondrial disorder
  * Severe liver disease other than hepatitis B or C due to interference with systemic cytokine production
  * Uncontrolled hypertension defined as resting systolic blood pressure (BP) >180 mmHg or diastolic BP >100 mmHg
  * Indicators of unstable ischemic heart disease
  * New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, uncontrolled angina, or uncontrolled arrhythmia
  * Pulmonary disease requiring the use of supplemental oxygen
  * Active malignancy (excluding non-melanoma skin cancers) within 24 weeks prior to enrollment
  * Surgery/trauma/injury/fracture within 12 weeks prior to enrollment that may limit ability to perform physical function testing.
  * Acute infection (skin infection, sinus infection, uncomplicated upper respiratory infection, dental infection, etc) within 2 weeks of study entry will be excluded until the infection has resolved for at least 2 weeks
  * Chronic, deeper infections (complicated pneumonia, bone infection, liver abscess, deep wound infection, etc) must have completed treatment and show no evidence of ongoing infection for at least 12 weeks
  * History of stroke with residual deficits
  * Any medical condition that does not allow for a non-contrasted MRI study (ie, pacemaker, shrapnel, other devices or hardware)
  * AIDS-defining opportunistic infection75 within the 24 weeks prior to enrollment
  * Severe anemia, defined as a hemoglobin of 9 mg/dL or less
  * Participants on anticoagulants (clopidogrel, Coumadin, etc). Patients on short-acting anticoagulant therapy requiring dose cessation for only 48-72 hours can be considered for muscle biopsy with approval by their treating physician.
  * Aspirin and Non-steroidal anti-inflammatory agents are not exclusions but should be stopped 1 week prior to biopsy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected participants will be those living with HIV, between the ages of 50-75 years, recruited from the University of Colorado Infectious Diseases Group Practice HIV-uninfected participants were previous enrolled and completed an IRB approved protocol (historical database).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
ADP/ATP measurement (mitochondrial function) | At Baseline
  ADP/ATP ratio between HIV-infected and uninfected subjects

SECONDARY OUTCOMES:
Protein citrate synthase | At Baseline
  Total protein citrate synthase between HIV-infected and seronegative subjects
Respiratory control ratio (RCR) | At Baseline
  Respiratory control ratio (RCR) between HIV-infected and uninfected subjects
Inflammatory markers | At Baseline
  Relationship between markers of inflammation (final panel to be determined, but most likely sTNFR1 and 2 in addition to multiplex panel of IL-6, IL-10, CRP, IFN-G) and their effect on mitochondrial function
Muscle function | At Baseline
  Relationship between measures of muscle function (strength, physical function) and mitochondrial function
TDF to TAF change | At Baseline
  A separate group of participants changing from TDF-based ART to TAF-based ART will also have mitochondrial function measures before and after change. The inclusion criteria are similar except the age range is 18-70.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
IPD is kept private per UC Denver restrictions